CLINICAL TRIAL: NCT00486226
Title: The SUNRISE Registry - A Multicenter Post-Market Surveillance With the CORDIS ENTERPRISE™ Vascular Reconstruction Device and Delivery System
Brief Title: The Registry to Study Safety and Performance of the CORDIS Vascular Reconstruction Device and Delivery System
Acronym: SUNRISE
Status: Completed | Type: Observational
Sponsor: Codman & Shurtleff (Industry)
Responsible Party: Sponsor
Other Study IDs: EN07-01
Record Dates: First submitted 2007-06-13; First posted 2007-06-14 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1 Endovascular: All patients implanted with an CORDIS ENTERPRISE Vascular Reconstruction Device.
  Interventions: Device: Vascular Reconstruction Device

INTERVENTIONS:
Device: Vascular Reconstruction Device — CORDIS ENTERPRISE™ VRD
  Other Names: ENTERPRISE; Codman ENTERPRISE; Codman VRD

SUMMARY:
The objective of the registry is to evaluate the real world safety and performance of the CORDIS ENTERPRISE™ Vascular Reconstruction Device and Delivery System (VRD) to facilitate endovascular coil embolization of intracranial aneurysms.

DETAILED DESCRIPTION:
The data will be collected in consecutive subjects treated with the commercially available product and following standard clinical practice. This registry will be limited to subjects who have received only the CORDIS ENTERPRISE™ VRD during the index procedure. While only limited inclusion or exclusion criteria are specified, uniform, complete and accurate data will be collected peri-procedurally, during the index hospitalization, and during follow-up up to 6 months. All subjects should be treated according to the Instruction For Use (IFU) including conduct of the VRD placement, coiling procedure, application of antiplatelet medication and any other medical therapy to be provided according to local usual practice.

ELIGIBILITY:
Inclusion Criteria:

* The subject must be >= 18 years of age and less than 80 years.
* Diagnosis of a ruptured (Hunt and Hess Grade I - III) or unruptured intracranial aneurysm at the time of the treatment
* Subject (or his/her legal representative) provides written informed consent for the use of his/her peri-procedural and follow-up data

Exclusion Criteria:

* Diagnosis of Hunt and Hess Grade IV or V subarachnoid hemorrhage at the time of the treatment
* Severe co-morbidity associated with a life-expectancy of less than six months
* Poor neurological status at baseline
* Known allergies to Nitinol metal
* Known allergies to aspirin, heparin, ticlopidine, or clopidogrel or unable or unwilling to tolerate therapy
* Participation in an investigational drug or another device study is only allowed after written approval of the coordinating investigator or Cordis Medical Monitor.
* Implantation of an intracranial stent associated with the symptomatic distribution within 12 weeks prior to the index procedure
* Implantation of carotid stent associated with the symptomatic distribution within 12 weeks prior to the index procedure
* Atrial fibrillation or known cardiac disorders likely to be associated with cardioembolic symptoms.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering of an intracranial aneurysm and necessitating an endovascular treatment.
  Patients who meet all of the general inclusion criteria and none of the exclusion criteria and who agree to voluntarily sign a informed consent form will be enrolled into the study.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2007-06-01 (Actual); Primary Completion 2012-12-01 (Actual); Study Completion 2013-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bendszus Martin, MD, Principal Investigator — Wuerzburg University Hospital; Boris Lubicz, MD, Principal Investigator — Université Libre de Bruxelles
Locations (1):
- Université Libre de Bruxelles, Brussels, Belgium

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 Endovascular: All patients implanted with an CORDIS ENTERPRISE Vascular Reconstruction Device (VRD). Vascular Reconstruction Device: CORDIS ENTERPRISE™ VRD
Period: Overall Study
Arm/Group | 1 Endovascular
Started | 105
Completed | 92
Not Completed | 13
Not completed — Death | 3
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 8

BASELINE CHARACTERISTICS:
Groups:
- 1 Endovascular: All patients implanted with an CORDIS ENTERPRISE Vascular Reconstruction Device and were consented before the procedure. Vascular Reconstruction Device: CORDIS ENTERPRISE™ VRD
Arm/Group | 1 Endovascular
Number analyzed (Participants) | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75
  Male | 30
Medical History [Number; unit: Participants]
  Cardiovascular Disease | 4
  Chronic Pulmonary Disease | 1
  Immunologic | 1
  Endocrice/Metabolic Disease | 1
  Diabetes | 2
  Renal Disease | 2
  Cancer | 6
  Dyslipidemia/Hypercolesterolemia | 4
  Vasculitis | 1
  Obesity | 1
  Smoking | 1
  Other | 4
  Hypertension | 38
Neurological History [Number; unit: Participants]
  Recurrent Headache | 18
  Epilepsy | 3
  Cranial Nerve Palsy/ Paresis | 2
  TIA/CVA | 21
Previous Neurological Surgical Procedures [Count of Participants; unit: Participants] | 36

OUTCOME MEASURES:

1. Primary Outcome: The Successful Intracranial VRD Placement With Satisfactory Coil Mass Position Without the Occurrence of Any Device and/or Procedure Related Serious Adverse Event (SAE)
Description: Successful intracranial VRD placement is defined as stable VRD placement with complete coverage of the aneurysm neck and parent artery patency. Satisfactory coil mass position is defined as VRD maintains coil position within the sac with parent artery patency as defined angiographically
Time Frame: Intra-procedure
Measure: Number (95% Confidence Interval); unit: participants
Groups:
- 1 Endovascular: All patients implanted with an CORDIS ENTERPRISE Vascular Reconstruction Device who signed consent before the procedure. Vascular Reconstruction Device: CORDIS ENTERPRISE™ VRD
Arm/Group | 1 Endovascular
Number analyzed (Participants) | 105
participants | 64 [51.6 to 70.0]

2. Secondary Outcome: Device or Procedure Related Adverse Events (AEs)
Description: Incidence of device or procedure related adverse events during the index procedure and till discharge
Time Frame: index procedure to discharge; an average of 3.8 days
Measure: Number; unit: participants
Groups:
- 1 Endovascular: All patients implanted with an CORDIS ENTERPRISE Vascular Reconstruction Device. Vascular Reconstruction Device: CORDIS ENTERPRISE™ VRD
Arm/Group | 1 Endovascular
Number analyzed (Participants) | 105
participants | 14

3. Secondary Outcome: Satisfactory Coil Mass Position
Description: Satisfactory coil mass position is defined as VRD maintains coil position within the sac with parent artery patency as defined angiographically
Time Frame: 6 months
Population: no data was available for 33 subjects; either because the investigator didn't submit the images or due to poor quality of the submitted images
Measure: Number; unit: participants
Arm/Group | 1 Endovascular
Number analyzed (Participants) | 72
participants | 60

4. Secondary Outcome: Aneurysm Occlusion
Description: Aneurysm occlusion was assessed using the Raymond Scale (Class 1 - Complete Obliteration / Class 2 - Residual Neck / Class 3 - Residual Aneurysm)
Time Frame: post procedure to 6 months
Population: no data was available for 21 subjects post-procedure and 26 subjects at 6 months follow-up; either because the investigator didn't submit the images or due to poor quality of the submitted images
Measure: Number; unit: participants
Groups:
- Endovascular - Occlusion Results Immediately Post-procedure: Aneurysm occlusion was assessed immediately post procedure using the Raymond Scale.
- Endovascular - Occlusion Results at 6 Months Follow-up: Aneurysm occlusion assessed at 6 months follow-up using the Raymond Scale.
Arm/Group | Endovascular - Occlusion Results Immediately Post-procedure | Endovascular - Occlusion Results at 6 Months Follow-up
Number analyzed (Participants) | 84 | 79
participants
  Complete Occlusion (Raymond 1) | 17 | 46
  Neck Remnant (Raymond 2) | 19 | 8
  Residual Aneurysm (Raymond 3) | 48 | 25

ADVERSE EVENTS:
Time Frame: procedure until 6 months follow-up
Description: At each evaluation of a subject enrolled in the registry (procedure, discharge, 6 months follow-up) the investigator determined whether any adverse events had occurred.
Arm/Group | 1 Endovascular
Serious Adverse Events (participants affected / at risk) | 5/105
Other Adverse Events (participants affected / at risk) | 21/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Endovascular (N=105)
Ischemic Stroke (Nervous system disorders) | 1 (1) — Ischemic Stroke in a different territory than the stented one
retroperitoneal hematoma (Injury, poisoning and procedural complications) | 1 (1) — retroperitoneal hematoma requiring additional hospitalization
Thrombophlebitis (Vascular disorders) | 1 (1) — Left superior limb thrombophlebitis and atrial fibrillation Headache and right hemiparesis
stent thrombosis (Injury, poisoning and procedural complications) | 1 (1) — Incomplete stent thrombosis started after stent and first coil placement.
Cancer (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Lung metastasis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Endovascular (N=105)
stent thrombosis (Injury, poisoning and procedural complications) | 2 (2)
embolization/ re-embolization of non-study aneurysm (Nervous system disorders) | 5 (7)
coil protrusion (Injury, poisoning and procedural complications) | 5 (5) — In four subjects coil protrusion occurred before placement of the Enterprise stent and was hence not related to the device. In the remaining subject the timing of coil protrusion (before/after stent placement) was not specified by the investigator.
stent migration (Injury, poisoning and procedural complications) | 2 (2)
cholangitis with septicemia (Hepatobiliary disorders) | 1 (1) — moderate sclerosing cholangitis post cholecystectomy and septicemia
stretched/unravelled coil (Injury, poisoning and procedural complications) | 2 (2)
perforator infarction (Nervous system disorders) | 1 (1)
subdural hematoma (Nervous system disorders) | 1 (1)
visual disturbances with cintilating scotoma (Nervous system disorders) | 1 (1)
Phasic Disorders (Musculoskeletal and connective tissue disorders) | 1 (1)
temporo-spatial disorientation (Nervous system disorders) | 1 (1)
Epistaxis (Injury, poisoning and procedural complications) | 1 (1)
Headache (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was powered to have a total of 250 subjects, but was stopped early due to slow enrollment. Hence, this study ended up having only 105 total subjects, making it underpowered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No